CLINICAL TRIAL: NCT06215820
Title: A Multi-Center, Randomized, Double-Blind, Placebo- (Double-Dummy) and Active-Controlled, Parallel-Group Study of MR-107A-02 for the Treatment of Acute Postoperative Pain Following Bunionectomy
Brief Title: Study of MR-107A-02 for the Treatment of Acute Postoperative Pain Following Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Viatris Specialty LLC (Industry)
Collaborators: Mylan Specialty, LP (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR-107A-02-TFZ-3001
Record Dates: First submitted 2023-12-22; First posted 2024-01-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Acute Pain; Post Operative Pain; Pain
Keywords: Pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Pain | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MR-107A-02 (Experimental): 15 mg Twice daily (BID) during in patient phase (0-48 hours following randomization) 15 mg BID dosing morning and evening, during out patient phase (5 days) .
  Interventions: Drug: MR-107A-02; Procedure: Bunionectomy
- Tramadol (Active Comparator): 50 mg, administered every 6 hours (q6h) during the in patient phase (0-48 hours following randomization).
  Placebo will be administered during out patient phase.
  Interventions: Drug: Tramadol; Drug: Placebo; Procedure: Bunionectomy
- Placebo (Placebo Comparator): Placebo is administered every 6 hours (q6h) during the in patient phase (0-48 hours following randomization) and twice daily during the out patient phase.
  Interventions: Drug: Placebo; Procedure: Bunionectomy

INTERVENTIONS:
Drug: MR-107A-02 — tablet
  Arms: MR-107A-02
Drug: Tramadol — over-encapsulated tablet
  Arms: Tramadol
Drug: Placebo — over-encapsulated tablet and/or tablet
  Arms: Placebo; Tramadol
Procedure: Bunionectomy — Primary unilateral bunionectomy with first metatarsal osteotomy under regional anesthesia

SUMMARY:
MR-107A-02 is being studied to investigate its efficacy and safety for treatment of acute pain after bunionectomy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Requirement for a primary unilateral bunionectomy
2. Has an American Society of Anesthesiologists Physical Status of I, II, or III.
3. Pain Intensity (PI) using a Numeric Rating Scale (NRS-R) ≥4 at any given timepoint during the 9 hours after removal of the popliteal sciatic block
4. Rating of moderate or severe pain on a 4-point categorical pain rating scale (i.e., none, mild, moderate, severe) during the 9 hours after removal of the popliteal sciatic block
5. Able to understand and complete the study requirements (including literacy, to enable diary and questionnaire completion), provide written informed consent, and agree to abide by the study protocol and its restrictions.

Key Exclusion Criteria:

1. Previously dosed with this formulation of MR-107A-02.
2. Subjects with a contralateral foot bunionectomy in the past 6 months.
3. Subject has a concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain that is not strictly related to the bunionectomy, and which may confound the postoperative assessments.
4. Known hypersensitivity to aspirin, NSAIDs or other medication used in the study.
5. Body mass index (BMI) >40 kg/m2 at screening.
6. Body weight of <43 kg at screening.
7. History of GI bleeding or peptic ulcer disease.
8. Known active inflammatory bowel disease, e.g., Crohn's Disease or ulcerative colitis.
9. A history of bleeding disorders that may affect coagulation.
10. Subjects with prior stroke or transient ischemic attack in the past 12 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference (SPID) for MR-107A-02 versus placebo. | 48 hours after randomization
  SPID based on a 0 to 10-point numeric rating scale at rest (NRS-R) for MR-107A-02 versus placebo.

SECONDARY OUTCOMES:
Number of doses of opioid rescue medication taken for MR-107A-02 versus placebo. | 7 days after randomization
  Number of doses of opioid rescue medication over the combined in-patient and outpatient treatment phases MR-107A-02 versus placebo.
Proportion of subjects using no opioid rescue medication MR-107A-02 versus placebo. | 7 days after randomization
  Proportion of subjects using no opioid rescue medication over the combined in-patient and outpatient treatment phases MR-107A-02 versus placebo.

OTHER OUTCOMES:
Summed Pain Intensity Difference (SPID) for tramadol versus placebo. | 48 hours after randomization
  SPID based on a 0 to 10-point numeric rating scale at rest (NRS-R) for tramadol versus placebo.
Summed Pain Intensity Difference (SPID) for MR-107A-02 versus tramadol | 48 hours after randomization
  SPID based on a 0 to 10-point numeric rating scale at rest (NRS-R) for MR-107A-02 versus tramadol.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Vogt, Study Director — Viatris Inc.
Locations (15):
- United States (15):
  - Investigator site 114, Sheffield, Alabama
  - Investigator site 115, Phoenix, Arizona
  - Investigator site 103, Anaheim, California
  - Investigator site 110, Riverside, California
  - Investigator site 112, Miami, Florida
  - Investigator site 108, Tampa, Florida
  - Investigator site 109, Atlanta, Georgia
  - Investigator site 104, O'Fallon, Illinois
  - Investigator site 102, Pasadena, Maryland
  - Investigator site 113, Bellaire, Texas
  - Investigator site 107, Carrollton, Texas
  - Investigator site 106, Houston, Texas
  - Investigator site 111, McAllen, Texas
  - Investigator site 105, San Antonio, Texas
  - Investigator site 101, Salt Lake City, Utah